CLINICAL TRIAL: NCT02504736
Title: 24 Week Open Label, Single Arm Study of Colesevelam in High Risk South Asians With Suboptimal LDL-c Levels Despite Maximally Tolerated Statin Therapy
Brief Title: Colesevelam, Lipids And Sugars, South Asian Canadian Trial
Acronym: CLASS-ACT
Status: Completed | Type: Observational
Sponsor: Canadian Collaborative Research Network (Other)
Collaborators: Valeant Canada Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CLASS ACT-24-FEB-2015
Record Dates: First submitted 2015-07-13; First posted 2015-07-22 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Dyslipidemia
Keywords: LDL cholesterol; A1c; High risk South Asians; Colesevelam
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the effect of colesevelam on LDL levels and A1c in high-risk , dysglycemic South Asians (with diabetes, and/or with CAD and concomitant metabolic syndrome) whose LDL remains above target despite optimal statin use.

DETAILED DESCRIPTION:
This is a prospective, non-controlled, open label, multicenter trial of colesevelam in Canadian South Asian adults at high cardiovascular risk.

1. 15-20 clinical sites from Ontario, Quebec, Manitoba and British Columbia will be selected from CCRN's network of primary care physicians and cardiologists to identify patients having stable type 2 diabetes or documented stable CAD with metabolic syndrome who are on maximally tolerated statin therapy, with LDL >2.0 mmol/L or non-HDL > 2.6 mmol/L.
2. Following informed consent, patients will be screened at baseline for HbA1c, fasting blood glucose, lipid profile, renal function and liver enzymes.
3. Baseline demographics, CAD and diabetes documentation and concurrent drug therapy will be collected.
4. 250 eligible patients will receive a physician prescription of colesevelam (Lodalis) 625 mg tablets (3 tablets taken twice daily) for 24 weeks.
5. Physicians will be requested not to change lipid or diabetes therapy over the 24 week course of the trial.
6. Patients will be contacted at 2 and 12 weeks (visit 3 and 4) via a phone call to assess adherence to the prescribed therapy, review other concurrent medications and assess for any adverse events.
7. The week 24 visit (study visit 5) will include collection of fasting blood work as per screening visit, review of concurrent drug therapy and a final assessment for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Individuals of South Asian ethnicity; self-declared, at least 3 of 4 grandparents born in a South Asian country (i.e. India, Pakistan, Bangladesh, Sri Lanka, Nepal and Bhutan)
* Either Diabetes, or Coronary artery disease with metabolic syndrome
* Currently receiving maximally tolerated dose of statin therapy (at least Atorvastatin 20 mg or Rosuvastatin 10 mg)
* LDL >2.0 mmol/L or non-HDL >2.6 mmol/L
* Patient is willing to provide written consent
* Age ≥ 18 years

Exclusion Criteria:

* Receiving lipid-lowering agents, other than statins or ezetimibe
* Any changes made to current lipid lowering therapy in the last 12 weeks
* Uncontrolled diabetes (HbA1c >0.10)
* TG > 5.0 mmol/L
* Significant hepatic or renal disease (ALT > 2x ULN or eGFR < 30 mL/min/1.73 m²)
* Ongoing participation in any randomized clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals of South Asian ethnicity; self-declared, at least 3 of 4 grandparents born in a South Asian country (i.e. India, Pakistan, Bangladesh, Sri Lanka, Nepal and Bhutan)
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
The % difference in LDL between baseline and end of study | 6 months

SECONDARY OUTCOMES:
The % change in HbA1c levels between baseline and end of study | 6 months
The absolute change in LDL and non-HDL levels between baseline and end of study | 6 months
The safety and tolerability of colesevelam will be determined by the patient reported side/adverse effects and/or hospitalization related to Colesevelam. The side effects will be captured at Visit 3, 4 and 5. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Milan K Gupta, MD, Principal Investigator — McMaster University, Hamilton, ON Canada; University of Toronto, Toronto, ON Canada; Narendra Singh, MD, Principal Investigator — Georgia Regents University, Georgia, US
Locations (1):
- Dr. Milan Gupta,MD, Brampton, Ontario, Canada

REFERENCES:
- [Background] Corsini A, Windler E, Farnier M. Colesevelam hydrochloride: usefulness of a specifically engineered bile acid sequestrant for lowering LDL-cholesterol. Eur J Cardiovasc Prev Rehabil. 2009 Feb;16(1):1-9. doi: 10.1097/HJR.0b013e32831215db. PMID 19237992
- [Background] Aggarwal S, Loomba RS, Arora RR. Efficacy of colesevelam on lowering glycemia and lipids. J Cardiovasc Pharmacol. 2012 Feb;59(2):198-205. doi: 10.1097/FJC.0b013e31823a109f. PMID 21983746
- [Background] Goldberg RB. Improving glycemic and cholesterol control through an integrated approach incorporating colesevelam - a clinical perspective. Diabetes Metab Syndr Obes. 2009 May 5;2:11-21. doi: 10.2147/dmsott.s3866. PMID 21437115
- [Background] Brunetti L, DeSantis EH. Patient tolerance and acceptance of colesevelam hydrochloride: focus on type-2 diabetes mellitus. P T. 2015 Jan;40(1):62-7. PMID 25628509
- [Background] Jialal I, Abby SL, Misir S, Nagendran S. Concomitant reduction in low-density lipoprotein cholesterol and glycated hemoglobin with colesevelam hydrochloride in patients with type 2 diabetes: a pooled analysis. Metab Syndr Relat Disord. 2009 Jun;7(3):255-8. doi: 10.1089/met.2009.0007. PMID 19344229
- [Background] Fonseca VA, Rosenstock J, Wang AC, Truitt KE, Jones MR. Colesevelam HCl improves glycemic control and reduces LDL cholesterol in patients with inadequately controlled type 2 diabetes on sulfonylurea-based therapy. Diabetes Care. 2008 Aug;31(8):1479-84. doi: 10.2337/dc08-0283. Epub 2008 May 5. PMID 18458145
- [Background] Zieve FJ, Kalin MF, Schwartz SL, Jones MR, Bailey WL. Results of the glucose-lowering effect of WelChol study (GLOWS): a randomized, double-blind, placebo-controlled pilot study evaluating the effect of colesevelam hydrochloride on glycemic control in subjects with type 2 diabetes. Clin Ther. 2007 Jan;29(1):74-83. doi: 10.1016/j.clinthera.2007.01.003. PMID 17379048